CLINICAL TRIAL: NCT05831124
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND STUDY OF THE SAFETY AND IMMUNOGENICITY OF A MULTIVALENT PNEUMOCOCCAL CONJUGATE VACCINE WITH AN ADJUVANT ADMINISTERED IN ADULTS 50 THROUGH 64 YEARS OF AGE
Brief Title: A Study to Learn About a Type of Pneumococcal Vaccine With a New Ingredient (PF-07872411) Intended to Enhance the Effects of the Vaccine Which is Given to Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4941001
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low dose multivalent pneumococcal conjugate vaccine formulation A (Experimental): Stage 1 - Participants will be randomized to receive a single injection.
  Interventions: Other: Low dose multivalent pneumococcal conjugate vaccine formulation A
- Low dose multivalent pneumococcal conjugate vaccine formulation B (Experimental): Stage 2 - Participants will be randomized to receive a single injection.
  Interventions: Other: Low dose multivalent pneumococcal conjugate vaccine formulation B
- Low dose of multivalent pneumococcal conjugate vaccine control (Active Comparator): Primary control - Stages 1 and 2 - Participants will be randomized to receive a single injection.
  Interventions: Biological: Low dose of multivalent pneumococcal conjugate vaccine control
- Standard dose multivalent pneumococcal conjugate vaccine control (Active Comparator): Control - Stages 1 and 2 - Participants will be randomized to receive a single injection.
  Interventions: Biological: Standard dose multivalent pneumococcal conjugate vaccine control

INTERVENTIONS:
Other: Low dose multivalent pneumococcal conjugate vaccine formulation A — Biological
  Arms: Low dose multivalent pneumococcal conjugate vaccine formulation A
Other: Low dose multivalent pneumococcal conjugate vaccine formulation B — Biological
  Arms: Low dose multivalent pneumococcal conjugate vaccine formulation B
Biological: Low dose of multivalent pneumococcal conjugate vaccine control — low dose multivalent pneumococcal conjugate vaccine
  Other Names: Primary control
  Arms: Low dose of multivalent pneumococcal conjugate vaccine control
Biological: Standard dose multivalent pneumococcal conjugate vaccine control — multivalent pneumococcal conjugate vaccine
  Other Names: Control
  Arms: Standard dose multivalent pneumococcal conjugate vaccine control

SUMMARY:
The purpose of this clinical trial is to learn about a pneumococcal vaccine with a new ingredient (PF-07872411) intended to enhance the effects of the vaccine. This pneumococcal vaccine with the new ingredient may prevent the diseases caused by pneumococcal bacteria like meningitis, sepsis, ear infections and sinusitis.

Meningitis is an infection in which the tissue around the brain and spine is swollen.

Sepsis is a very serious infection in your blood caused by a germ (a bacteria). Sinusitis is when your sinuses (the air-filled spaces inside your nose and head), are infected.

This study is seeking for healthy participants who:

* are above 50 years of age and less than 64 years of age.
* have not taken any vaccine for pneumococcal diseases before.
* have not taken any vaccines with additional ingredients within 1 year before administration of the study vaccine.

All participants will receive a single study vaccine shot in the upper arm muscle at the study clinic. The study will compare the experiences of people receiving the vaccine with a new ingredient in the vaccine to those without the new ingredient. This will be done by comparing 2 different dose levels of the new ingredient. It will also be compared against people who receive the vaccine without the new ingredient and at different dose levels. This will help the study team establish if the vaccine with a new ingredient is safe and effective.

Participants will take part in this study for about 12 months. During this time participants will have up to 6 clinic visits. At these clinic visits, participants will be asked if any side effects were experienced. The participants will also have to give blood samples during these visits.

Some participants will need to have blood taken for laboratory tests before they can be judged to be eligible to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥50 and ≤64 years of age at the time of consent.
* Adults determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study, including those with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease, within 6 months before receipt of study intervention.
* Female participants of childbearing potential or male participants able to father children and who are willing to use acceptable methods of contraception for at least 28 days after the last dose of study intervention; or female participants not of childbearing potential; or male participants not able to father children.

Exclusion Criteria:

* History of a severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component in pneumococcal conjugate vaccines and any other diphtheria toxoid-containing vaccine.
* Serious chronic disorder, including history of metastatic malignancy, severe COPD requiring supplemental oxygen, end-stage renal disease with or without dialysis, cirrhosis of the liver, clinically unstable cardiac disease, or any other disorder, that in the investigator's opinion, would make the participant inappropriate for entry into the study.
* History of microbiologically proven invasive disease caused by S pneumoniae.
* Current febrile illness (body temperature ≥100.4°F [≥38.0°C]) or other acute illness within 48 hours before study intervention administration.
* Pregnant female participants or breastfeeding female participants (known or suspected).
* Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt of any licensed or investigational pneumococcal vaccine through study participation.
* Receipt of any inactivated or otherwise nonlive vaccine within 14 days or any live vaccine within 28 days before administration of study intervention.
* Receipt of an adjuvanted vaccine containing QS-21 (or similar saponin adjuvant), MPL, or MF59 within 1 year before administration of study intervention

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting local reactions within 7 days after vaccination | 7 days
  Local reactions (redness, swelling, pain at the injection site) after vaccination.
Percentage of participants reporting systemic events within 7 days after vaccination | 7 days
  Systemic events (fever, vomiting, diarrhea, headache, fatigue, chills, muscle pain, and joint pain) after vaccination.
Percentage of participants reporting Adverse Events (AEs) within 1 month after vaccination | 1 month
  Adverse Events occurring within 1 month after vaccination.
Percentage of participants reporting Serious Adverse Events (SAEs) within 6 months after vaccination | 6 months
  SAEs occurring within 6 months after vaccination.
Percentage of participants reporting Serious Adverse Events (SAEs) withing 12 months after vaccination | 12 months
  SAEs occurring within 12 months after vaccination.
Percentage of participants reporting Newly Diagnosed Chronic Medical Conditions (NDCMCs) within 6 months after vaccination | 6 months
  NDCMCs occurring within 6 months after vaccination.
Percentage of participants reporting Newly Diagnosed Chronic Medical Conditions (NDCMCs) withing 12 months after vaccination | 12 months
  NDCMCs occurring within 12 months after vaccination.
Percentage of participants reporting Medically Attended Adverse Events (MAAEs) within 6 months after vaccination | 6 months
  MAAEs occurring within 6 months after vaccination.
Percentage of participants reporting Medically Attended Adverse Events (MAAEs) within 12 months after vaccination | 12 months
  MAAEs occurring within 12 months after vaccination.
Stage 1 and Stage 2 Only - Percentage of participants with abnormal hematology and chemistry laboratory values 2 weeks after vaccination | 2 weeks
  Abnormal hematology and chemistry laboratory values occurring 2 weeks after vaccination.

SECONDARY OUTCOMES:
Pneumococcal opsonophagocytic activity (OPA) titers | 1 month
  OPA geometric mean titers (GMTs) 1 month after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Research Centers of America, Hollywood, Florida
  - Centennial Medical Group, Columbia, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Rochester Clinical Research, LLC, Rochester, New York
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4941001